CLINICAL TRIAL: NCT07242482
Title: Study on the Clinical Value of Circulating Immune Markers in Prognostic Evaluation of Postoperative Lung Cancer Patients
Brief Title: Circulating Immune Markers for Prognostic Evaluation in Postoperative Lung Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Zhao Jun (Other)
Responsible Party: Sponsor-Investigator, Zhao Jun, Thoracic Surgery, The First Affiliated Hospital of Soochow University
Organization: The First Affiliated Hospital of Soochow University (Other)
Other Study IDs: 2025979
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer (Diagnosis); Biomarkers / Blood
Keywords: Peripheral Blood; Tumor antigen specific T cells; Teff/Treg ratio; Prognostic Evaluation
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Preoperative Peripheral Blood Immune Marker Analysis. — Preoperative collection of approximately 5 mL peripheral blood via venipuncture, followed by isolation of peripheral blood mononuclear cells (PBMCs) using Ficoll density gradient centrifugation. PBMCs are analyzed via multiparametric flow cytometry on a BD FACSCanto II system to quantify antigen-specific effector T cells (ETASTs, co-expressing CD137 and IFN-γ after ex vivo stimulation with NSCLC antigen peptide pools like NY-ESO-1 and MAGE-A3) and the effector T cell to regulatory T cell ratio (Teff/Treg, with Teff as CD4+/CD8+ expressing IFN-γ/TNF-α/IL-2 and Treg as CD4+CD25+FoxP3+). Analysis uses FlowJo software, targeting 100,000 events per sample. This non-invasive prognostic assessment is distinct from routine clinical blood tests by its focus on tumor-specific immune activation and balance, without therapeutic intent or alteration of standard care.

SUMMARY:
Investigating the Clinical Value of Tumor Antigen-Specific T Cells and Immune Cell Balance in Peripheral Blood of Non-Small Cell Lung Cancer Patients for Prognostic Evaluation.

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) remains the leading cause of cancer-related mortality worldwide, with surgical resection serving as the curative approach for early to intermediate stages. However, postoperative recurrence rates are high in stages IB (with high-risk features such as tumor >4 cm, poor differentiation, visceral pleural invasion, vascular invasion, or wedge resection) to IIIB, necessitating improved prognostic tools beyond TNM staging to optimize adjuvant therapies like chemotherapy or immunotherapy.

This study investigates peripheral blood immune markers as non-invasive prognostic indicators. Antigen-specific effector T cells (ETASTs) are identified via multiparametric flow cytometry, co-expressing CD137 (a T-cell activation marker) and IFN-γ (an effector cytokine) following ex vivo stimulation with tumor-associated antigens. The effector T cell to regulatory T cell ratio (Teff/Treg) reflects systemic immune homeostasis, with imbalances promoting tumor immune evasion.

Blood samples (approximately 10 mL) are collected preoperatively via venipuncture and processed within 4 hours. Peripheral blood mononuclear cells (PBMCs) are isolated using Ficoll density gradient centrifugation. For ETAST detection, PBMCs undergo stimulation with a peptide pool of common NSCLC antigens (e.g., NY-ESO-1, MAGE-A3) for 6 hours in the presence of brefeldin A, followed by intracellular staining and analysis on a BD FACSCanto II flow cytometer. Teff cells are defined as CD4+ or CD8+ T cells expressing IFN-γ, TNF-α, or IL-2; Treg cells as CD4+CD25+FoxP3+. Data acquisition targets at least 100,000 events per sample, with analysis using FlowJo software.

Follow-up includes clinical assessments every 3 months for the first 2 years, then every 6 months up to 3 years, monitoring recurrence via CT scans, PET-CT if indicated, and survival endpoints. Exploratory analyses may incorporate next-generation sequencing for driver mutations (e.g., EGFR, ALK) from tumor tissue to correlate with immune profiles.

Ethical considerations prioritize participant safety, with all procedures approved by the institutional review board. Data are de-identified and stored securely, complying with GCP standards.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years.
* Diagnosed with primary non-small cell lung cancer (NSCLC) and scheduled to undergo curative lung resection at the Department of Thoracic Surgery of our institution.
* Postoperative pathological stage is IB (with tumor size >4cm or high-risk factors: poor differentiation, vascular invasion, visceral pleural invasion, sub-lobar resection, etc.), IIA, IIB, or IIIB (according to the AJCC 8th edition).
* ECOG performance status of 0 or 1.
* Voluntarily signs the informed consent form.

Exclusion Criteria:

* Received any neoadjuvant therapy prior to surgery.
* History of other active malignancies.
* Diagnosed with severe autoimmune diseases, active infections, or immunodeficiency disorders.
* Presence of severe cardiac, hepatic, or renal dysfunction.
* Pregnant or lactating women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a single-center, prospective, observational cohort study. The study population consists of adult patients (18-80 years) with primary non-small cell lung cancer who are scheduled for curative resection at the Thoracic Surgery Department. Eligible patients must have a postoperative pathological stage of IB (with high-risk features), IIA, IIB, or IIIB (AJCC 8th ed.), an ECOG status of 0-1, and provide informed consent. Key exclusions include prior neoadjuvant therapy, other active cancers, and significant comorbidities. A total of 200 participants are planned to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-17 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence-Free Survival | 3 years postoperatively
  The time from the date of surgery to the first occurrence of disease recurrence, metastasis, or death from any cause.

SECONDARY OUTCOMES:
Overall Survival | 3 years postoperatively
  The time from the date of surgery to death from any cause.
Correlation between immune markers and clinicopathological features | Baseline (preoperative)
  To analyze the associations between preoperative levels of ETASTs, Teff/Treg ratio, and clinicopathological characteristics such as TNM stage, pathological type, and driver gene mutation status.
Immunological prognostic scoring model (Nomogram) | 3 years postoperatively
  To develop a nomogram model integrating significant immune markers (e.g., ETASTs, Teff/Treg ratio) and clinical variables (e.g., TNM stage) for predicting recurrence-free survival. The model will be internally validated using the Bootstrap method, and its discrimination (C-index) and calibration will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Soochow university, Suzhou, Jiangsu 215000, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided